CLINICAL TRIAL: NCT07364890
Title: Platelet-Derived Growth Factors to Enhance Healing and Reduce Post-Extraction Complications in Smokers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Amal Jamjoom, BDS, MS., Assistant Professor at KAU, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 120-11-24
Record Dates: First submitted 2025-12-13; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Smoke Exposure
Keywords: Smokers; A- PRF; Extraction; Socket

STUDY DESIGN:
Intervention Model Description: One extraction socket receives A-PRF and the contralateral side will act a a control.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A- PRF in Extraction sockets in smokers (Experimental): A- PRF in Extraction sockets in smokers.
  Interventions: Drug: A- PRF
- Control (No Intervention): Control site will not receive anything

INTERVENTIONS:
Drug: A- PRF — A-PRF will be placed in one extraction socket
  Other Names: Advanced Platelet Rich Fibrin
  Arms: A- PRF in Extraction sockets in smokers

SUMMARY:
This study is a randomized controlled clinical trial with a split-mouth design to evaluate the effect of Advanced Platelet-Rich Fibrin (A-PRF) application on socket healing following dental extractions in smokers. In the split-mouth design, each participant serves as their own control, minimizing inter-subject variability and controlling for potential confounders such as smoking habits, oral hygiene, and systemic health conditions.

Bilateral tooth extractions will be performed for each participant, with one extraction site randomly assigned to receive socket preservation using an A-PRF plug, while the contralateral site will be left to heal naturally without intervention.

The study will be conducted at the Faculty of Dentistry and the University Dental Hospital, King Abdulaziz University, Jeddah, Saudi Arabia. Recruitment began in December 2025 and will continue until the targeted sample size is achieved.

DETAILED DESCRIPTION:
Participants will be recruited using a convenience sampling approach from the College of Dentistry and the University Dental Hospital at King Abdulaziz University, Jeddah, Saudi Arabia.

Patients requiring bilateral tooth extractions and initially appearing eligible based on their medical records will be identified. Eligibility will be further confirmed through direct interviews to verify smoking habits (≥10 cigarettes per day) and to ensure compliance with the inclusion and exclusion criteria.

Patients who meet the eligibility requirements will be informed about the nature and purpose of the study, and those who agree to participate will provide written informed consent.

Following recruitment, each participant will have one extraction site randomly assigned to receive A-PRF treatment (intervention), while the contralateral site will serve as the control, according to a split-mouth design. Recruitment will commence in January 2026 and will continue until the planned sample size is achieved. Here is the **fully converted future-tense version**, polished and suitable for a **study protocol / PRS / methods section**:

All dental extractions will be performed by a periodontist under local anesthesia (2% lidocaine with 1:100,000 epinephrine) using simple atraumatic techniques to preserve the socket architecture and minimize trauma to the surrounding soft and hard tissues. No surgical extractions will be performed.

A-PRF will be prepared immediately after tooth extraction. Intravenous blood samples will be collected from each participant using sterile glass-coated 9-mL tubes without an anticoagulant. The blood samples will be processed immediately by centrifugation at 1300 rpm for 14 minutes to obtain Advanced Platelet-Rich Fibrin (A-PRF).

Following centrifugation, the fibrin clots will be carefully separated from the red blood cell layer, transferred to a PRF box, and gently compressed into plugs.

At the intervention sites, the prepared A-PRF plugs will be gently adapted into the extraction socket immediately after tooth removal and stabilized using a figure-of-eight suture to secure the material and protect the healing site. At the control sites, no A-PRF will be placed; only a figure-of-eight suture will be applied to stabilize the blood clot and support natural healing.

Standard postoperative instructions will be provided to all participants to promote optimal healing and minimize postoperative complications.

Intraoral digital scans will be performed to assess soft-tissue healing immediately after extraction and at 7 and 14 days post-extraction. Participants will also be asked to complete a patient-reported experience questionnaire at one week and again at the time of suture removal (two weeks post-extraction).

ELIGIBILITY:
Inclusion Criteria:

* Smokers
* Aged 18 years or older
* Actively smoking at least 10 cigarettes per day
* Requiring bilateral extractions.

Exclusion Criteria:

* Patients younger than 18 years
* Diabetes mellitus
* Hypertension
* Bleeding disorders
* Pregnant or lactating women
* Individuals who used tobacco products other than conventional cigarettes (such as e-cigarettes or waterpipes) were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Socket size using intra-oral scan | 3 weeks
  Socket size will be measured using intra-oral digital scanning. Three-dimensional scans of the extraction site will be obtained and analyzed using digital software to delineate socket margins and calculate the socket surface area (mm²).

CONTACTS AND LOCATIONS:
Overall Officials: Amal G Jamjoom, MS, Principal Investigator — King Abdulaziz University
Locations (1):
- King AbdulAziz University, Jeddah, Mekkah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in publications arising from this study will be shared. This will include demographic variables, smoking status, clinical outcomes related to soft tissue healing, intraoral scan measurements, and patient-reported outcome questionnaire data. No identifiable information will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: PD will be available beginning 6 months after publication of the primary results and will remain available for up to 5 years thereafter.
Access Criteria: Access to de-identified individual participant data will be granted to qualified researchers who submit a scientifically sound proposal outlining the research objectives and planned analyses. Requests will be reviewed by the principal investigator to ensure alignment with the original study aims, ethical approval, and data protection requirements. Approved applicants will be required to sign a data use agreement prior to data release. Data will be provided in a secure, de-identified format and used solely for the approved purpose.

REFERENCES:
- [Background] Yerke LM, Jamjoom A, Zahid TM, Cohen RE. The Effect of Platelet-Rich Fibrin, Calcium Sulfate Hemihydrate, Platelet-Rich Plasma and Resorbable Collagen on Soft Tissue Closure of Extraction Sites. J Funct Biomater. 2017 May 25;8(2):17. doi: 10.3390/jfb8020017. PMID 28587096
- [Background] Pan J, Xu Q, Hou J, Wu Y, Liu Y, Li R, Pan Y, Zhang D. Effect of platelet-rich fibrin on alveolar ridge preservation: A systematic review. J Am Dent Assoc. 2019 Sep;150(9):766-778. doi: 10.1016/j.adaj.2019.04.025. PMID 31439204
- [Background] Malcangi G, Patano A, Palmieri G, Di Pede C, Latini G, Inchingolo AD, Hazballa D, de Ruvo E, Garofoli G, Inchingolo F, Dipalma G, Minetti E, Inchingolo AM. Maxillary Sinus Augmentation Using Autologous Platelet Concentrates (Platelet-Rich Plasma, Platelet-Rich Fibrin, and Concentrated Growth Factor) Combined with Bone Graft: A Systematic Review. Cells. 2023 Jul 6;12(13):1797. doi: 10.3390/cells12131797. PMID 37443831
- [Background] El Bagdadi K, Kubesch A, Yu X, Al-Maawi S, Orlowska A, Dias A, Booms P, Dohle E, Sader R, Kirkpatrick CJ, Choukroun J, Ghanaati S. Reduction of relative centrifugal forces increases growth factor release within solid platelet-rich-fibrin (PRF)-based matrices: a proof of concept of LSCC (low speed centrifugation concept). Eur J Trauma Emerg Surg. 2019 Jun;45(3):467-479. doi: 10.1007/s00068-017-0785-7. Epub 2017 Mar 21. PMID 28324162
- [Background] Choukroun J, Diss A, Simonpieri A, Girard MO, Schoeffler C, Dohan SL, Dohan AJ, Mouhyi J, Dohan DM. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part IV: clinical effects on tissue healing. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e56-60. doi: 10.1016/j.tripleo.2005.07.011. PMID 16504852
- [Background] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part II: platelet-related biologic features. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e45-50. doi: 10.1016/j.tripleo.2005.07.009. Epub 2006 Jan 10. PMID 16504850
- [Background] Dohan Ehrenfest DM, Rasmusson L, Albrektsson T. Classification of platelet concentrates: from pure platelet-rich plasma (P-PRP) to leucocyte- and platelet-rich fibrin (L-PRF). Trends Biotechnol. 2009 Mar;27(3):158-67. doi: 10.1016/j.tibtech.2008.11.009. Epub 2009 Jan 31. PMID 19187989
- [Background] Dohan Ehrenfest DM, Del Corso M, Diss A, Mouhyi J, Charrier JB. Three-dimensional architecture and cell composition of a Choukroun's platelet-rich fibrin clot and membrane. J Periodontol. 2010 Apr;81(4):546-55. doi: 10.1902/jop.2009.090531. PMID 20373539
- [Background] Alshehri, A., et al., Assessment of the low-speed centrifugation concept modified in the release of fibroblast growth factor-2 in Saudi healthy patient. Saudi Journal of Oral Sciences, 2020. 7(3): p. 169-173.
- [Background] Fujioka-Kobayashi M, Miron RJ, Hernandez M, Kandalam U, Zhang Y, Choukroun J. Optimized Platelet-Rich Fibrin With the Low-Speed Concept: Growth Factor Release, Biocompatibility, and Cellular Response. J Periodontol. 2017 Jan;88(1):112-121. doi: 10.1902/jop.2016.160443. Epub 2016 Sep 2. PMID 27587367
- [Background] Lalla E, Papapanou PN. Diabetes mellitus and periodontitis: a tale of two common interrelated diseases. Nat Rev Endocrinol. 2011 Jun 28;7(12):738-48. doi: 10.1038/nrendo.2011.106. PMID 21709707
- [Background] Souto-Maior JR, Pellizzer EP, de Luna Gomes JM, Dds CAAL, Dds JFSJ, Vasconcelos BCDE, de Moraes SLD. Influence of Diabetes on the Survival Rate and Marginal Bone Loss of Dental Implants: An Overview of Systematic Reviews. J Oral Implantol. 2019 Aug;45(4):334-340. doi: 10.1563/aaid-joi-D-19-00087. Epub 2019 May 1. PMID 31042455
- [Background] Mealey BL, Ocampo GL. Diabetes mellitus and periodontal disease. Periodontol 2000. 2007;44:127-53. doi: 10.1111/j.1600-0757.2006.00193.x. No abstract available. PMID 17474930
- [Background] De Angelis P, Manicone PF, Gasparini G, De Filippis I, Liguori MG, De Angelis S, Cannata F, D'Addona A. The Effect of Controlled Diabetes and Hyperglycemia on Implant Placement with Simultaneous Horizontal Guided Bone Regeneration: A Clinical Retrospective Analysis. Biomed Res Int. 2021 Jun 14;2021:9931505. doi: 10.1155/2021/9931505. eCollection 2021. PMID 34222488
- [Background] Power DJ, Sambrook PJ, Goss AN. The healing of dental extraction sockets in insulin-dependent diabetic patients: a prospective controlled observational study. Aust Dent J. 2019 Mar;64(1):111-116. doi: 10.1111/adj.12669. Epub 2019 Jan 2. PMID 30525221
- [Background] Huang S, Dang H, Huynh W, Sambrook PJ, Goss AN. The healing of dental extraction sockets in patients with Type 2 diabetes on oral hypoglycaemics: a prospective cohort. Aust Dent J. 2013 Mar;58(1):89-93. doi: 10.1111/adj.12029. Epub 2013 Jan 28. PMID 23441797
- [Background] Aronovich S, Skope LW, Kelly JP, Kyriakides TC. The relationship of glycemic control to the outcomes of dental extractions. J Oral Maxillofac Surg. 2010 Dec;68(12):2955-61. doi: 10.1016/j.joms.2010.05.006. Epub 2010 Oct 14. PMID 20950911
- [Background] Gadicherla S, Smriti K, Roy S, Pentapati KC, Rajan J, Walia A. Comparison of Extraction Socket Healing in Non-Diabetic, Prediabetic, and Type 2 Diabetic Patients. Clin Cosmet Investig Dent. 2020 Jul 20;12:291-296. doi: 10.2147/CCIDE.S264196. eCollection 2020. PMID 32765113
- [Background] Shen X, Shen X, Li B, Zhu W, Fu Y, Xu R, Du Y, Cheng J, Jiang H. Abnormal macrophage polarization impedes the healing of diabetes-associated tooth sockets. Bone. 2021 Feb;143:115618. doi: 10.1016/j.bone.2020.115618. Epub 2020 Aug 26. PMID 32858254
- [Background] Devlin H, Sloan P. Early bone healing events in the human extraction socket. Int J Oral Maxillofac Surg. 2002 Dec;31(6):641-5. doi: 10.1054/ijom.2002.0292. PMID 12521322
- [Background] de Sousa Gomes P, Daugela P, Poskevicius L, Mariano L, Fernandes MH. Molecular and Cellular Aspects of Socket Healing in the Absence and Presence of Graft Materials and Autologous Platelet Concentrates: a Focused Review. J Oral Maxillofac Res. 2019 Sep 5;10(3):e2. doi: 10.5037/jomr.2019.10302. eCollection 2019 Jul-Sep. PMID 31620264
- [Background] Zhou S, Li G, Zhou T, Zhang S, Xue H, Geng J, Liu W, Sun Y. The role of IFT140 in early bone healing of tooth extraction sockets. Oral Dis. 2022 May;28(4):1188-1197. doi: 10.1111/odi.13833. Epub 2021 Mar 16. PMID 33682229
- [Background] Wang Q, Liu J, Qi S, Liao X, Liu D, Pan J. Clinical analysis of medication related osteonecrosis of the jaws: A growing severe complication in China. J Dent Sci. 2018 Sep;13(3):190-197. doi: 10.1016/j.jds.2017.12.003. Epub 2018 Feb 6. PMID 30895120
- [Background] Yoo JJ, Kim DW, Kim MY, Kim YT, Yoon JH. The effect of diabetes on tooth loss caused by periodontal disease: A nationwide population-based cohort study in South Korea. J Periodontol. 2019 Jun;90(6):576-583. doi: 10.1002/JPER.18-0480. Epub 2019 Mar 12. PMID 30548930
- [Background] Al-Rubeaan K, Al Derwish M, Ouizi S, Youssef AM, Subhani SN, Ibrahim HM, Alamri BN. Diabetic foot complications and their risk factors from a large retrospective cohort study. PLoS One. 2015 May 6;10(5):e0124446. doi: 10.1371/journal.pone.0124446. eCollection 2015. PMID 25946144
- [Background] Singh N, Armstrong DG, Lipsky BA. Preventing foot ulcers in patients with diabetes. JAMA. 2005 Jan 12;293(2):217-28. doi: 10.1001/jama.293.2.217. PMID 15644549
- [Background] Davis VL, Abukabda AB, Radio NM, Witt-Enderby PA, Clafshenkel WP, Cairone JV, Rutkowski JL. Platelet-rich preparations to improve healing. Part I: workable options for every size practice. J Oral Implantol. 2014 Aug;40(4):500-10. doi: 10.1563/AAID-JOI-D-12-00104. PMID 25106016
- [Background] Mohseni Homagarani Y, Adlparvar K, Teimuri S, Tarrahi MJ, Nilchian F. The effect of diabetes mellitus on oral health-related quality of life: A systematic review and meta-analysis study. Front Public Health. 2023 Feb 24;11:1112008. doi: 10.3389/fpubh.2023.1112008. eCollection 2023. PMID 36908413
- [Background] Kudiyirickal MG, Pappachan JM. Diabetes mellitus and oral health. Endocrine. 2015 May;49(1):27-34. doi: 10.1007/s12020-014-0496-3. Epub 2014 Dec 9. PMID 25487035
- [Background] Alwin Robert A, Al Dawish MA. Microvascular complications among patients with diabetes: An emerging health problem in Saudi Arabia. Diab Vasc Dis Res. 2019 May;16(3):227-235. doi: 10.1177/1479164118820714. Epub 2019 Jan 1. PMID 30599757

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT07364890/Prot_SAP_000.pdf